CLINICAL TRIAL: NCT03821350
Title: The Effect of Comorbid Psychiatric Disorders and Information Leaflet on Results of Transforaminal Epidural Steroid Injection
Brief Title: The Effect of Comorbid Psychiatric Conditions on Results of Transforaminal Epidural Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Yeliz Bahar Ozdemir, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2014.0089
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain; Radiculopathy
Keywords: Transforaminal epidural steroid injection; Radicular pain
MeSH Terms: conditions — Low Back Pain; Radiculopathy

STUDY DESIGN:
Intervention Model Description: Parallel group
Who Masked: Investigator
Masking Description: The study was designed as prospective, single blinded, randomized controlled study. Patients were randomized into two groups. The enrollment of the participants was carried out by an independent researcher. Pre and post-injection evaluation was performed by the investigators who had no knowledge about the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group was given verbal information
- Leaflet Group (Experimental): The second group was given verbal information and a detailed information leaflet with written and visual content
  Interventions: Other: Information leaflet

INTERVENTIONS:
Other: Information leaflet — The written and visual information form prepared specifically for the patients was aimed to provide detailed information by clearly expressing the procedure, the suggestions that will be needed before and after injection (what to bring next, what circumstances may not be done, the control visit day after the procedure etc.) to be applied on before the injection day.
  Arms: Leaflet Group

SUMMARY:
Low back pain (LBP) and radiculopathic pain are a major socio-economic problem affecting all age groups. 70% of people consult a doctor at least once in their life due to LBP. Radicular pain is thought to be caused by inflammation of the spinal nerve roots near the intervertebral disc injury. In this context, fluoroscopic guided transforaminal epidural steroid injection (TFESI) has been increasingly preferred in patients who can not benefit from conservative approach in the treatment of lumbosacral radiculopathic pain due to lumbar disc herniation in recent years.

The assessment of comorbid psychiatric conditions such as depression, anxiety, and somatization disorder and given the detailed and visual information to patients who will be undergone TFESI could affect the result of the treatment in a good way. The pain questionnaire used for objectively evaluating injection outcomes is personality dependent and there are many factors that can affect it.

DETAILED DESCRIPTION:
Although information leaflets given to patients prior to surgical or non-surgical interventions have not yet been used as a standard in each clinic, the effects on patients have been frequently researched in recently. A detailed description of the treatment, the devices to be used and the disclosure of the steps of the procedure may have an effect on the result of the treatment. The aim of the study; (1) the presence of comorbid psychiatric conditions in patients with lumbar disc hernia and radiculopathy, (2) to evaluate the effect of the written and visual informative form given before the injection of the lumbosacral TFESI.

ELIGIBILITY:
Inclusion Criteria:

* lumbar radiculopathy due to lumbar disc herniation,
* unresponsive to conservative treatments,
* duration of pain is less than 3 months,
* patients scheduled for the first time with TFESI.

Exclusion Criteria:

* the cases when fluoroscopy or epidural injection is contraindicated (coagulation disorders, pregnancy etc...),
* underwent epidural injection in the last 6 months,
* to have a history of lumbar spinal surgery,
* inflammatory diseases (rheumatoid arthritis, spondyloarthropathy),
* spinal infection or malignancy,
* to benefit from six-week medical treatment,
* be reluctant to participate in the work and follow up,
* who are illiterate,
* the patients with psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2015-12-25 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale | 3 months
  The patient is asked to give a score between 1 and 10 to explain the pain level.
Oswestry disability index | 3 months
  The oswestry disability index is a survey designed to investigate how lumbar and leg pain affects their daily lives. It consists of 10 questions investigating the general life activity of the patient. The patient receives at least 0 points and at most 5 points from each question. The higher scores indicate that increased disability.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 3 months
  The Hospital Anxiety and Depression Scale is an easy-to-use questionnaire consisting of 14 questions that examines the symptoms of depression with 7 questions and anxiety with 7 questions.
Somatosensory Amplification Scale | 3 months
  The Somatosensory Amplification Scale is a scale consisting of 10 items. The items include a series of disturbing bodily sensations that do not present a disease.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coudeyre E, Poiraudeau S, Revel M, Kahan A, Drape JL, Ravaud P. Beneficial effects of information leaflets before spinal steroid injection. Joint Bone Spine. 2002 Dec;69(6):597-603. doi: 10.1016/s1297-319x(02)00457-8. PMID 12537268
- [Background] Sivaganesan A, Chotai S, Parker SL, Asher AL, McGirt MJ, Devin CJ. Predictors of the efficacy of epidural steroid injections for structural lumbar degenerative pathology. Spine J. 2016 Aug;16(8):928-34. doi: 10.1016/j.spinee.2015.11.058. Epub 2015 Dec 9. PMID 26689476